CLINICAL TRIAL: NCT04646278
Title: Estimation of Coronary Artery Hemodynamic Profiles Using Cineangiography Technique
Brief Title: Coronary Hemodynamics by Coronary Angiography
Acronym: ESCARGOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KangWon National University Hospital (Other)
Collaborators: The Korean Society of Cardiology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B-2017-01-012-015
Record Dates: First submitted 2020-11-04; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; Index of microcirculatory resistance; TIMI frame count; Fractional flow reserve; Coronary flow reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients who underwent coronary angiography and further hyperemic stimui
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyperemic stimuli (Experimental): Hyperemic stimuli of coronary flow by adenosine or nicorandil injection
  Interventions: Drug: Hyperemic stimuli

INTERVENTIONS:
Drug: Hyperemic stimuli — Hyperemic simuli of coronary flow by adenosine or nicorandil injection
  Other Names: Hyperemia

SUMMARY:
Study for developing techniques to evaluate coronary artery hemodynamic profiles by conventional angiography without more dedicated measuring devices.

DETAILED DESCRIPTION:
* Methods: Compare TIMI frame count, coronary clearance frame count in baseline/hyperemic coronary angiography with FFR, CFR, IMR and derive correlation, receiver-operating characteristic curve to find new tools estimating coronary hemodynamics by conventional angiography only.

A TIMI frame count is measured by counting the angiographic image cine frames during a head of radiocontrast column runs from the entry of left anterior descending artery (LAD) to the distal end.

A coronary clearance frame count is measured by counting the angiographic image cine frames during a tail of radiocontrast column runs from the entry of LAD to the distal end.

Baseline angiography is performed without any stimulation and hyperemic angiography is performed after intracoronary injection of adenosine 300ug or nicorandiol 2mg.

Inclusion criteria

* Patient who underwent physiologic study using a pressure wire for intermediate coronary lesion after coronary angiography

Exclusion criteria

* ST elevation myocardial infarction
* Cardiogenic shock
* Congestive heart failure with pulmonary edema
* LVEF < 30%
* Previous history of coronary revascularization
* Chronic total occlusion
* 3 vessel disease
* Target lesion at distal segments or branches

ELIGIBILITY:
Inclusion criteria

* Patient who underwent physiologic study using a pressure wire for intermediate coronary lesion after coronary angiography

Exclusion criteria

* ST elevation myocardial infarction
* Cardiogenic shock
* Congestive heart failure with pulmonary edema
* LVEF < 30%
* Previous history of coronary revascularization
* Chronic total occlusion
* 3 vessel disease
* Target lesion at distal segments or branches

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
TIMI frame count | Imediately after the procedure
  frame count between the beginning and end of contrast column head
Coronary Clearance Frame Count | Imediately after the procedure
  frame count between the beginning and end of contrast column tail
Index of microcirculatory resistance | During the procedure
  derived from distal coronary pressure by transit time

SECONDARY OUTCOMES:
Fractional flow reserve | During the procedure
  measured by pressure wire
Coronary flow reserve | During the procedure
  measured by pressure wire by thermodilution technique

CONTACTS AND LOCATIONS:
Overall Officials: Bong-Ki Lee, MD, PhD, Principal Investigator — KangWon National University Hospital
Locations (1):
- Kangwon National University Hospital, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Could be shared after necessary discussions
Supporting Information: Study Protocol
Time Frame: after publication
Access Criteria: Investigator who I permitted